CLINICAL TRIAL: NCT05245630
Title: Comparison of Real-time Robotic Arm-assisted 18F-FDG PET/CT-guided Lung Biopsy Versus PET Fused CT- Fluoroscopy-guided Lung Biopsy: a Randomized Trial to Assess Diagnostic Performance and Patient Safety.
Brief Title: Comparison of Robotic Arm-assisted PET/CT-guided Lung Biopsy With PET Fused CT- Fluoroscopy-guided Lung Biopsy
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/6832/MD/594
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Lung Diseases; Adenocarcinoma of Lung
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic arm assisted PET/CT guided biopsy: In this group, participants were recruited for robotic-assisted PET/CT guided biopsy from the FDG avid lung lesions.
  biopsies were done using an automated robotic arm (MAXIO-EX, Perfint healthcare Pvt Ltd, Chennai, India) to guide the needle for biopsy. It is a robotic arm with a four-ax guide arm and a planning console. Pre-interventional fused PET/CT images from Biograph mCT 16 scanner were sent via LAN cable to the device (MAXIO-EX) console.
  Interventions: Procedure: Robotic arm assisted PET/CT guided biopsy; Procedure: PET fused CT-Fluoroscopy guided biopsy
- PET fused CT-Fluoroscopy guided biopsy: In this group, participants were recruited for PET fused CT-Fluoroscopy guided biopsy from the FDG avid lung lesions.
  A biopsy needle was placed to the target lesion on PET/CT under CT fluoroscopy
  Interventions: Procedure: Robotic arm assisted PET/CT guided biopsy; Procedure: PET fused CT-Fluoroscopy guided biopsy

INTERVENTIONS:
Procedure: Robotic arm assisted PET/CT guided biopsy — After preparing the participant for the procedure, the participant was positioned on the PET/CT table with the immobilizer.
  An automated robotic arm (MAXIO-EX, Perfint healthcare Pvt Ltd, Chennai, India) was used to guide the needle for biopsy.
  Co-axial 18 G biopsy needle (BARD Biopsy disposable coaxial biopsy needle pack, Bard Peripheral Vascular, Inc., Arizona, USA) was inserted according to the orientation planned by the robotic biopsy device.
  After the location is ensured, the trocar stylet is removed from the coaxial cannula and specimens were retrieved using a semiautomated biopsy gun.
  A repeat CT chest was acquired two hours after the procedure to rule out post-procedural complications.
  Complications during the procedure were noted, and immediate management was done.
Procedure: PET fused CT-Fluoroscopy guided biopsy — CT fluoroscopy was used to place the biopsy needle to the FDG avid lung lesion

SUMMARY:
Patients with suspicious lung lesions were undertaken for PET/CT directed under CT fluoroscopy lung biopsy or robotic-assisted biopsy. The biopsy planning including patient positioning was done after F18-FDG PET/CT whole body or regional imaging of the patient. Written consent was obtained and the patient will be prepared for the biopsy. Lung biopsies were done using a semi-automatic biopsy gun under the imaging guidance (PET fused CT fluoroscopy) following aseptic precautions. Follow-up CT scans were taken post-biopsy. The time consumed for the procedure, radiation exposure to the interventionist, complications and diagnostic yield in both the arms were compared.

DETAILED DESCRIPTION:
Patients with clinical suspicion of lung lesions were recruited for FDG PET/CT. Based on the PET/CT findings and clinical details a PET/CT guided biopsy was planned. The patients were assigned to the two arms. In the first arm, participants underwent a robotic-assisted biopsy. In the second arm, participants underwent PET/CT-directed CT fluoroscopy-guided lung biopsy. The biopsy planning including patient positioning was done after F18-FDG PET/CT whole body or regional imaging of the patient. Written consent was obtained and the patient will be prepared for the biopsy. Lung biopsies were done using a semi-automatic biopsy gun under the imaging guidance (PET fused CT fluoroscopy) following aseptic precautions. Follow-up CT scans were taken post-biopsy. The time consumed for the procedure, radiation exposure to the interventionist, complications and diagnostic yield in both the arms were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. FDG avid amenable lung lesion
3. INR < 1.2 and Platelet counts > 80,000/mm3

Exclusion Criteria:

1. Participants with pre-existing bleeding diathesis like hemophilia, coagulopathy defined by INR ≥ 1.2 and Platelet counts ≤ 80,000/mm3
2. Participants who refuse to provide the written informed consent
3. Signs of hypoperfusion like cyanosis, hypotension etc.
4. Presence of hypoxemia (SpO2 < 95% -measured in a pulse oximeter)
5. Pregnant/Lactating females participants
6. Non-cooperative participants
7. Inaccessible lesions (based on the decision made on pre-biopsy planning)
8. CoVID-19 positive participants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants attending the pulmonary medicine department with clinical suspicion of lung lesions were referred to the Department of Nuclear Medicine for lung biopsies were recruited for the study. The participants were randomly assigned to either of the two intervention arms. Baseline heart rate, blood pressure, oxygen saturation and respiratory system examination were done for all the participants included in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
To compare the accuracy ( in percentage) of trans-thoracic percutaneous PET fused CT-fluoroscopy guided lung biopsy and automated robotic arm assisted PET/CT guided lung biopsy | three months
  Histology reports of the biopsies were recorded and the mutation analysis,
  Adequacy of the sample was decided by the pathologist who received the sample and when inadequate, we were notified accordingly by the Department of Pathology.
  The histopathological results were analyzed. True positive, True negative False-positive and False-negative were calculated for both the groups.
  The diagnostic accuracy in percentage for both arms will be calculated and compared.

SECONDARY OUTCOMES:
To compare the radiation exposure and complication in the both arms | three months
  Procedure related complications and radiation exposure to the participants and interventionist were noted in the both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
Data generated or analyzed during the study are available from the primary investigator on a valuable and genuine request.